CLINICAL TRIAL: NCT03149328
Title: Electronic Patient-Reported Outcomes in Clinical Kidney Practice (ePRO Kidney)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Cambian Business Services, Inc. (Industry); Intogrey Research and Development Inc. (Industry); Alberta Health services (Other)
Responsible Party: Principal Investigator, Kara Schick-Makaroff, Principal Investigator, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00068365
Record Dates: First submitted 2017-05-01; First posted 2017-05-11 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Kidney Disease, End-Stage
Keywords: Home Dialysis; Person-Centred Care; Patient-Reported Outcome Measures; Process Evaluation; Educational Support; Electronic Patient-Reported Outcome Measures; Patient-Reported Experience Measures
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Training Support

STUDY DESIGN:
Intervention Model Description: Process evaluation with two phases (Phase 1: Usability Testing; Phase 2: Evaluation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Northern Alberta Renal Program (NARP) (Experimental): Provide in NARP (intervention group), 1) an electronic tool (ePRO) that facilitates real time PRO data collection and feedback in clinical practice, and 2) educational support to multidisciplinary home dialysis clinicians about how to use PROs routinely in their practice.
  Interventions: Other: Educational Support
- Southern Alberta Renal Program (SARP) (No Intervention): In SARP (comparator group), clinicians will not receive PRO feedback or education sessions.

INTERVENTIONS:
Other: Educational Support — In the intervention group, clinicians will be provided with PRO feedback for use in their clinical practice. They will also receive educational support on how to use PRO data at point of care.
  Arms: Northern Alberta Renal Program (NARP)

SUMMARY:
People living with end-stage kidney disease (ESKD) need dialysis or transplantation in order to stay alive. This illness and treatment significantly impact peoples' health, emotions, work and relationships. To promote person-centred care, healthcare professionals should be asking patients about what matters to them and using this feedback to plan and deliver care. Patient-reported outcome and experience questionnaires (jointly referred to as PROs) allow patients to provide information about their quality of life, symptoms and experiences with care. PROs are increasingly used to help healthcare professionals learn about what is important to patients and the impacts of illness or treatments from patients' point of view. Embedding feedback from patients into routine clinical practice is important in end-stage kidney disease because of the physical and quality of life challenges these patients face when living with kidney failure.

PROs provide vital and often missing information that the healthcare team can use to support patients. However, PROs administered via paper questionnaires have been perceived as cumbersome, difficult to integrate with other health information and do not provide immediate feedback.

In this research, home dialysis patients will have the opportunity to complete electronically administered PROs (ePROs) and healthcare professionals will receive education about how to use PRO information. The goal is to learn how to support healthcare professionals to routinely use this information to inform patient care, and see if this makes a difference in patients' symptoms, person-centred care, quality of life and satisfaction with care.

Learning what matters most to patients is essential for healthcare professionals to provide person-centred care. This research will address the gap in our understanding of how to best use patients' reports in healthcare. Findings of this research may ultimately improve the quality of healthcare for Canadians living with end-stage kidney disease.

DETAILED DESCRIPTION:
Objectives:

1. Understand the process of supporting clinicians to utilize PROs in multidisciplinary, home dialysis practice.
2. Examine to what extent utilization of PRO information is associated with differences in symptoms and person-centred care [primary outcomes], as well as satisfaction with care, utilization of health services, mental health, and QOL [secondary outcomes].

Approach:

To achieve these goals, a mixed methods design of process evaluation will be used to compare two groups: Northern and Southern Alberta Renal Programs, NARP (Edmonton) and SARP (Calgary). In Edmonton (Intervention group), patients and clinicians will be invited to participate in the study. Only patients will be invited to take part in the study in Calgary (Comparison group). The research study will be undertaken collaboratively with a Patient Advisory Committee and knowledge users.

Setting:

This research will be conducted among patients receiving home dialysis across Alberta Kidney Care, from its two units: Aberhart Clinic in the Northern Alberta Renal Program (NARP), and Sheldon M. Chumir Health Centre in the Southern Alberta Renal Program (SARP). NARP and SARP have 305 and 350 home dialysis patients respectively.

Methods:

The study is divided into two phases: Phase 1-Year 1 (Usability Testing) and Phase 2-Year 2 (Evaluation). SARP and NARP participants will be invited to complete ePROs for each of their scheduled appointments, every three months, throughout Phases 1 and 2.

Phase 1:

In NARP, the intervention group, interested patients will be approached and consent will be obtained. Before the clinic visit, the patient will complete a demographic survey, and the Edmonton Symptom Assessment Scale revised for renal patients (ESASr:Renal) using Cambian Navigator, a web-based ePRO system hosted by Cambian Business Services Inc. Survey results will be printed and given to the nurse, transcribed and placed in the patient' chart as well as on their electronic chart. NARP patients will also complete the Kidney Disease Quality of Life (KDQOL-36), the Patient Assessment of Care for Chronic Conditions (PACIC-20), and the EQ-5D-5L after their clinic appointment. These 3 outcome evaluation measures will not be included in patient charts, or be used by clinicians at point of care. Usability testing and formative evaluation with NARP patients will also include up to 5 focus groups and 10 interviews to discuss how they would like their PRO information to be used by clinicians. Usability testing and formative evaluation with NARP multidisciplinary clinicians will include a series of focus groups (3-4) to discuss the ideal process for ePROs surveys to be integrated in existing work structures. Findings from these focus groups will be used to refine the targeted workshops provided as an intervention in Phase 2.

In SARP, the comparator group, all patients meeting inclusion criteria will be invited to complete the consent form, demographic survey, and the ePRO survey tools collected in NARP, but not to participate in focus groups and interviews. The ePRO surveys will not be seen by the clinicians, but they will be informed of the study.

Phase 2:

Using a prospective design, the workshops (intervention) will occur in NARP. Clinicians will receive ePRO feedback as well as targeted education about how to use PRO information. Workshops will be offered every 1.5 months over the 6-month intervention period. Evaluation survey feedback will be sought at the end of each workshop to tailor information to clinicians' needs. In NARP, patients will continue to complete the PRO surveys before and after their clinic appointments. If other PRO measures are requested by clinicians in Phase 1, these will be added to Phase 2 data collection. Additionally, clinicians will be invited to complete an anonymous ticky-box form every 2 weeks, indicating if they reviewed the PRO information, and changed their decision-making based on the PRO information. All NARP clinicians will also be invited to participate in 1 interview (n=20). They will be asked to share examples of how they have used PRO information in their practice, and the challenges, benefits and facilitators of integrating ePROs in practice. Patient participants will also be invited to take part in a focus group (n=6) or interview (n=6) to discuss how they see clinicians following up on their PRO information.

In SARP, clinicians will provide usual care. Clinicians will not receive PRO information or participate in workshops. Education will be provide to SARP clinicians following completion of the study, as a form of knowledge translation.

Quantitative Evaluation:

Descriptive methods and statistical tests will be used to examine the trajectories of outcome measures for patients in the comparator and intervention groups. The area under the curve (AUC) will be calculated for each trajectory during the period that the patient is participating to create a summary score. Analysis of covariance (ANCOVA) will be used as the method of analysis to compare AUC scores of outcomes of both groups while controlling for within- and between-group differences, such as comorbidities, gender, age and dialysis type.

Qualitative Evaluation:

Qualitative data from focus groups and interviews will be recorded, transcribed verbatim and analyzed using the methodology of interpretive description. NVIVO, a qualitative software system, will be used to create a filing system and coding database. The first focus group/interview transcript in each phase will be read and re-read to generate an initial codebook. The codebooks will be iteratively refined throughout the analysis. Codes will be categorized and analyzed thematically. Patient and clinician data will be analyzed separately. Differences between pre- and post-implementation in NARP will also be examined.

ELIGIBILITY:
Patient inclusion:

* home dialysis patients attending regularly scheduled appointments in Edmonton at the Aberhart Clinic (NARP) or in Calgary at the Sheldon M. Chumir Health Centre (SARP)
* ≥18 years old
* able to read and speak English
* can provide written informed consent
* if a patient changes dialysis modality, they can continue to participate

Clinician inclusion:

* all clinical staff working with home dialysis patients at the Aberhart clinic in Edmonton (NARP)
* study co-investigators/collaborators who are NARP clinicians may choose to participate

Patient exclusion criteria:

* visual impairment
* cannot read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Schick-Makaroff, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Sheldon M. Chumir Health Centre, Calgary, Alberta
  - Aberhart Centre, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of analysis, anonymous, quantitative data will be made available online indefinitely to the public on a database, such as Dataverse. Dataverse is a public repository and the University of Alberta provides the infrastructure support for sharing datasets. (See (http://dataverse.org/)
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication the data will be available indefinately
Access Criteria: Anyone with a dataverse account will have access to the data

REFERENCES:
- [Derived] Schick-Makaroff K, Klarenbach S, Kwon JY, Cohen SR, Czupryn J, Lee L, Pauly R, MacRae JM, Forde B, Sawatzky R. Electronic patient-reported outcomes in clinical kidney practice (ePRO Kidney): a process evaluation of educational support for clinicians. Ther Adv Chronic Dis. 2023 Jun 12;14:20406223231173624. doi: 10.1177/20406223231173624. eCollection 2023. PMID 37332391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who attended a home dialysis clinic in either the Aberhart Center in Edmonton (NARP), between August 28, 2017 & August 30, 2019 or the Sheldon M Chumir Health Center in Calgary (SARP), between October 5, 2017 & October 31, 2019 and who met the inclusion criteria were invited to participate in this study. Patients were excluded if they were under 18 years of age, could not read or speak English or could not provide informed consent.
Pre-assignment Details: Patients were recruited and placed into their arm based on the clinic they were attending - there was no random assignment. 51 participants were clinicians (48) and family caregivers (3), these 2 participants groups were not part of the trial portion of the study.
Groups:
- Clinician Support and Education Around Use of PROs in Home Dialysis Clinic: In this study arm home dialysis clinic patient participants completed Electronic Patient Reported Outcome Measures (ePRO) every three months, the ePRO results for the ESASr were given to the nurse and placed in the patient chart (paper and electronic). This process helps to facilitate real time Patient Reported Outcomes (PRO) data collection and feedback in clinical practice.
  Educational Training and Support was provided to the multidisciplinary home dialysis clinicians on how to use the results of the patient completed ePROs routinely in their practice to support ongoing patient care.
  Kidney Patient Population: Northern Alberta Renal Program (NARP)
- Usual Care: In this study arm home dialysis clinic patient participants completed Electronic Patient Reported Outcome Measures (ePROs) every 3 months for study comparison data but this information was not shared with the home dialysis clinic clinicians and the clinicians did not have access to participant's assessment responses.
  Kidney Patient Population: Southern Alberta Renal Program (SARP)
Period: Overall Study
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Started | 284 | 259
Completed | 200 | 213
Not Completed | 84 | 46
Not completed — Withdrawal by Subject | 30 | 26
Not completed — Changed Dialysis Modality | 18 | 1
Not completed — Transplant | 9 | 1
Not completed — Lost to Follow-up | 25 | 16
Not completed — Left Study Site | 1 | 2
Not completed — Language Barrier | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: In this study arm home dialysis clinic patient participants completed Electronic Patient Reported Outcome Measures (ePROs) every 3 months for study comparison data but this information was not shared with the home dialysis clinic clinicians and the clinciains did not have access to participant's assessment responses.
  Kidney Patient Population: Southern Alberta Renal Program (SARP)
- Total: Total of all reporting groups
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care | Total
Number analyzed (Participants) | 284 | 259 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants chose not to answer - missing data
  years
    number analyzed (Participants) | 282 | 259 | 541
    (all) | 55.4 (13.3) | 56.7 (14.2) | 56.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants chose to not answer - missing data
  Participants
    number analyzed (Participants) | 282 | 259 | 541
    Female | 97 | 88 | 185
    Male | 185 | 171 | 356
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Asian was categorized as SAsian, Chinese, Filipino, SEAsian, WAsian, and Japanese; Other = Arab, LatinAm, Eth_other; More than one race = White and Eth_other, White and Aboriginal, White, Aboriginal and Eth_other, White and LatinAm
  Participants
    Race/Ethnicity: Aboriginal | 23 | 9 | 32
    Race/Ethnicity: Asian | 42 | 62 | 104
    Race/Ethnicity: White | 196 | 159 | 355
    Race/Ethnicity: Black | 4 | 10 | 14
    Race/Ethnicity: Other | 14 | 6 | 20
    Race/Ethnicity: More than one race/ethnicity | 5 | 12 | 17
    Race/Ethnicity: Unknown or not reported | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants] — Population: 2 participants chose to not answer - missing data
  Participants
    number analyzed (Participants) | 283 | 258 | 541
    Retired | 77 | 95 | 172
    Unable to Work | 82 | 61 | 143
    Working | 89 | 76 | 165
    Other | 35 | 26 | 61
Highlest Level of Education [Count of Participants; unit: Participants] — Population: 2 participants chose to not answer - missing data
  Participants
    number analyzed (Participants) | 284 | 257 | 541
    Elementary School | 18 | 5 | 23
    High School Graduate | 95 | 67 | 162
    College / Trade Diploma | 101 | 113 | 214
    Undergraduate Degree | 40 | 50 | 90
    Graduate Degree | 25 | 18 | 43
    Other | 5 | 4 | 9
Type of Dialysis [Count of Participants; unit: Participants] — Population: 2 participants chose not to answer - missing data
  Participants
    number analyzed (Participants) | 282 | 259 | 541
    Peritoneal | 199 | 187 | 386
    Home Hemodialysis | 75 | 65 | 140
    Nocturnal | 6 | 5 | 11
    Other | 2 | 2 | 4
Diagnoses [Count of Participants; unit: Participants]
  Diabetes | 116 | 83 | 199
  Hypertension | 182 | 186 | 368
  Myocardial Infarction | 27 | 26 | 53
  Heart Disease | 39 | 26 | 65
  Stroke | 16 | 10 | 26
  Leg Amputation | 10 | 7 | 17
  Lung Disease | 8 | 15 | 23
  Liver Disease | 2 | 6 | 8
  Arthritis | 38 | 49 | 87
  Cancer | 22 | 13 | 35
  Lower Back Pain | 43 | 40 | 83
  Depression | 36 | 31 | 67
  Other | 28 | 33 | 61

OUTCOME MEASURES:

1. Primary Outcome: Symptoms - Trajectory of Change
Description: Assessed using the symptoms/problems domain of the Kidney Disease Quality of Life 36-Item Short Form Survey (KDQOL-36). The Symptoms/Problems domain has 12 items, each representing a symptom or side effect of kidney disease based on the past 4 weeks with 5 response items ranging from "Not Bothered at all = 100" to "Extremely Bothered = 0". Min Score = 0; Max score = 100. Higher score indicates better health.
Time Frame: Trajectories of up to 24 months from start of enrollment to study completion
Population: Intent to treat population (all participants assigned to Clinician Support and Education as well as Usual Care). Based on Imputed dataset.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Patient Reported Outcome Surveys
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 284 | 259
Number analyzed (Patient Reported Outcome Surveys) | 1196 | 1056
score on a scale | 77.2 (14.2) | 76.2 (15.1)
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; We will examine the trajectories of outcome measures for patients in the comparator and intervention groups. The area under the curve (AUC) will be calculated for each trajectory during the period that the patient is participating to create a summary score. Null Hypothesis is that both groups are the same; Test type: Equivalence — Based on a power analysis for an ANCOVA comparing 2 groups using the area under the curve approach, a total sample 459 (655 x 70% response rate) will provide 80% power to detect effect sizes (f2) of moderate magnitude at a statistical significance level of 0.05 (e.g., f2 ranging from 0.15 for 1 covariate to 0.19 for 10 covariates); p = 0.30, ANCOVA — Threshold for statistical significance was p=0.05

2. Primary Outcome: Person-centred Care - Trajectory of Change
Description: Assessed using the Patient Assessment of Care for Chronic Conditions (PACIC-20), a patient-reported experience measure on satisfaction with care over the past 6 months. The PACIC-20 is a 20-item survey based on five subscales: (1) patient activation, (2) delivery system design and decision support, (3) goal setting and tailoring, (4) problem-solving and contextual counselling, and (5) follow-up and coordination. Each item is rated on a five-point scale (from "Almost never = 0" to "Almost always = 5") and the subscale and total scores are based on average scores across items. Min score = 0; Max score = 5. Higher scores indicates higher quality of care.
Time Frame: Trajectories of up to 24 months from start of enrollment to study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Patient Reported Outcome Surveys
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 284 | 259
Number analyzed (Patient Reported Outcome Surveys) | 1196 | 1056
score on a scale | 3.4 (1.1) | 3.5 (1.0)
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; We will examine the trajectories of outcome measures for patients in the comparator and intervention groups. The area under the curve (AUC) will be calculated for each trajectory during the period that the patient is participating to create a summary score. Null Hypothesis = both groups are the same; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.28, ANCOVA

3. Secondary Outcome: Utilization of Health Services
Description: Assessed using health services data (i.e. average number of hospital admissions, trips to the emergency room) determined through SPOR Platform and Alberta Health Services electronic health records. Higher numbers indicates worse outcomes.
Time Frame: From study enrollment until completion (up to 24 months)
Population: Health data for 5 participants classified as intervention were not found in the Alberta Health Services Database
Measure: Mean (Standard Deviation); unit: number of occurances
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 279 | 259
number of occurances
  Hospitalizations | 1.99 (2.15) | 2.33 (2.52)
  Emergency Room Visits | 5.72 (7.28) | 4.53 (5.58)
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; Analysis of covariance (ANCOVA) will be used as the method of analysis to compare outcomes of both groups while controlling for within- and between-group differences, such as comorbidities, gender, age and dialysis type. ANCOVA is necessary to control for baseline and potential confounders. Null hypotheses = No difference between groups in the number of hospitalizations; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.22, ANCOVA — Threshold for statistical Significance was p = 0.05
Statistical Analysis 2: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; Analysis of covariance (ANCOVA) will be used as the method of analysis to compare outcomes of both groups while controlling for within- and between-group differences, such as comorbidities, gender, age and dialysis type. ANCOVA is necessary to control for baseline and potential confounders. Null hypotheses = No difference between groups in the number of emergency room visits; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.10, ANCOVA — Threshold for statistical Significance was p = 0.05

4. Secondary Outcome: Number of Participants Who Selected "1 - Excellent" on Satisfaction With Care
Description: Assessed using one item added to the end of the Patient Assessment of Care for Chronic Conditions 20 item questionnaire (PACIC-20) related to care received. This item is from the NHS Outpatient Survey (2011). (RateClin) related to care received on a Likert-type scale from Excellent = 1 to Very Poor = 6. Min = 1, max = 6. The number of patients who selected "1 - Excellent" was tabulated and compared between the two groups. The higher the number the more patients who felt the care provided to them was excellent.
Time Frame: Up to 24 months from start of enrollment to study completion
Population: as for outcome 1
Measure: Count of Units; unit: Patient Reported Outcome Surveys
Units Other Than Participants: Patient Reported Outcome Surveys
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 284 | 259
Number analyzed (Patient Reported Outcome Surveys) | 1196 | 1056
Patient Reported Outcome Surveys | 654 | 547
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; Analysis of covariance (ANCOVA) will be used as the method of analysis to compare outcomes of both groups while controlling for within- and between-group differences, such as comorbidities, gender, age and dialysis type. ANCOVA is necessary to control for baseline and potential confounders. Null hypotheses = No difference between groups; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.18, ANCOVA — Threshold for statistical significance p = 0.05

5. Secondary Outcome: Mental Health - Trajectory of Change
Description: Assessed using the SF-12 mental component summary (MCS) subscale in the Kidney Disease Quality of Life 36-item Short-Form Survey (KDQOL-36). The SF-12 uses 2 items (psychological distress and psychological well being) to measure the MCS score. The summary score is transformed using Canadian norm-based scoring. The scores ranged from 0 (worst health) to 100 (best health). The higher the score the better the mental health.
Time Frame: Trajectories of up to 24 months from start of enrollment to study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Patient Reported Outcome Surveys
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 284 | 259
Number analyzed (Patient Reported Outcome Surveys) | 1196 | 1056
score on a scale | 50.9 (8.4) | 51.0 (8.3)
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.79, ANCOVA — Threshold for statistical significance p = 0.05

6. Secondary Outcome: Quality of Life - Trajectory of Change
Description: Assessed using the Euro Quality of Life EQ-5D-5L. This assessment uses a descriptive system for health-related Quality of Life states in adults consisting of 5 dimensions; Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension is scored between 1 = indicating no problem and 5 = indicating unable to/extreme problems. An EQ-5D summary index is derived by applying a formula (the Canadian standard value set) that attaches values (weights) to each of the levels in each dimension. Index min= 0.0 max = 1.0. The higher the index the better the quality of life/state of health.
Time Frame: Trajectories of up to 24 months from start of enrollment to study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Patient Reported Outcome Surveys
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
Number analyzed (Participants) | 284 | 259
Number analyzed (Patient Reported Outcome Surveys) | 1196 | 1056
score on a scale | 0.772 (0.182) | 0.745 (0.196)
Statistical Analysis 1: Comparison: Clinician Support and Education Around Use of PROs in Home Dialysis Clinic vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — Threshold for statistical significance p = 0.05

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Clinician Support and Education Around Use of PROs in Home Dialysis Clinic | Usual Care
All-Cause Mortality (participants affected / at risk) | 23/284 | 12/259
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/259
Other Adverse Events (participants affected / at risk) | 0/284 | 0/259

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03149328/Prot_SAP_000.pdf